CLINICAL TRIAL: NCT01797055
Title: Dose Escalating Study to Evaluate Pharmacokinetics, Efficacy and Safety of Apotransferrin in Atransferrinemia Patients
Brief Title: Apotransferrin in Atransferrinemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD2009.04
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Congenital Atransferrinemia
Keywords: transferrin; anemia; iron overload
MeSH Terms: conditions — Congenital atransferrinemia; Anemia; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- human apotransferrin (Experimental): intravenous apotransferrin every 4-8 weeks
  Interventions: Drug: Human apotransferrin

INTERVENTIONS:
Drug: Human apotransferrin — intravenous infusion

SUMMARY:
Atransferrinemia is a very rare disorder, which is caused by a deficiency of the protein transferrin. No regular treatment is available for these patients. The objective of this study is to investigate the pharmacokinetics, efficacy and safety of Apotransferrin replacement therapy in atransferrinemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of atransferrinemia, defined as serum levels of transferrin below 40 mg/dl
* Informed consent

Exclusion Criteria:

* Known with allergic reactions against human plasma or plasma products
* Having detectable anti-immunoglobulin A antibodies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 15 year
  Hemoglobin within normal range
pharmacokinetics of transferrin | first infusion and year 3
  serum transferrin levels measured on several time points before and after infusion
iron overload in organs | 15 years
  Elimination of iron overload (liver, heart)

SECONDARY OUTCOMES:
Iron overload | 15 years
  Serum Ferritin within normal values
Hematocrit | 15 years
  Hematocrit within normal values
Erythrocytes | 15 years
  Erythrocytes within normal values

OTHER OUTCOMES:
transferrin levels | 15 years
  Effective transferrin levels
adverse drug reactions | 15 years
  number of adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Cristina R Diaz de Heredia Rubio, PhD, MD, Principal Investigator — Vall d'Hebron, Spain; Katja Moser, MD, Principal Investigator — klinikum Aschaffenburg, Germany; Raffaella Mariani, MD, PhD, Principal Investigator — AO San Gerardo Monza, Italy; Alberto Piperno, MD, PhD, Principal Investigator — AO San Gerardo Monza, Italy
Locations (3):
- Klinikum Aschaffenburg, Aschaffenburg, Germany
- AO San Gerardo, Monza, Italy
- Vall d'Hebron Hospital, Barcelona, Spain